CLINICAL TRIAL: NCT04269746
Title: Assessment Of Long Noncoding RNA CCAT1 Using Real Time -Polymerase Chain Reaction In Colorectal Cancer Patients
Brief Title: Assessment Of Long Noncoding RNA CCAT1 In Colorectal Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alyaa Abd El-Rasoul Sayed Refae, Assistant lecturer, Assiut University
Other Study IDs: CCAT1 in colorectal cancer
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: The control population comprised normal healthy individuals.
  Interventions: Diagnostic Test: CCAT1
- Precancerous group: patients with precancerous colorectal diseases
  Interventions: Diagnostic Test: CCAT1
- CRC group: patients with colorectal cancer
  Interventions: Diagnostic Test: CCAT1

INTERVENTIONS:
Diagnostic Test: CCAT1 — Long Non coding RNA

SUMMARY:
1. Evaluate the diagnostic value of long noncoding RNA (CCAT1) expression by RT-PCR in peripheral blood in colorectal cancer patients versus normal healthy control personal.
2. Evaluate the clinical utility of detecting long noncoding RNA (CCAT1) expression in diagnosis of colorectal cancer patients & its relation to tumor staging.
3. Evaluate the clinical utility of detecting long noncoding RNA (CCAT1) expression in precancerous colorectal diseases.
4. Compare long noncoding RNA (CCAT1) expression with traditional marker; carcinoembryonic antigen (CEA) and Carbohydrate antigen 19-9 (CA19-9) in diagnosis of colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most commonly diagnosed cancer and the fourth leading cause of cancer mortality worldwide. Colorectal cancer is the 7th commonest cancer in Egypt, representing 3.47% of male cancers and 3% of female cancers. Cancer metastasis in the liver, which develops in 50% of CRC patients, represents the major cause of death in those patients .

CRC can be easily cured with surgery, if it is discovered and diagnosed early. Although in the recent years much progress has been achieved in screening for cancer, the prognosis of colorectal cancer is still poor. Colonoscopy is the standard screening method to detect early CRC .

Moreover, the other CRC screening tests (such as sigmoidoscopy, fecaloccult blood test (FOBT), tumor markers, fecal immunochemical test (FIT) and radiologic tests) have low sensitivity and specificity or high cost . Therefore, there is a great need for non-invasive and accurate biomarkers for detection of CRC.

Focusing into the physiological risk factors, genetic alterations may result from external influences like chemicals, radiation as well as pathogens (viruses) that disrupt the genome stability. Besides extensive studies on DNA damages in cell cycle regulation, past few decades evident the role of non-coding RNAs (ncRNAs) in the context of tumor biology. The existence of non-protein coding RNAs was known over years, where biological functions of these RNAs have been uncovered by progressive investigations. Non-coding RNAs have further classifications, among which the functions of micro RNAs (miRNAs) have been thoroughly explored. Thus, the concentration on the other type of ncRNA, the long non-coding RNAs (lncRNAs), is a yet emerging field in the research of cancer biology. A fraction of the genome comprises these lncRNAs who are actually poorly translated as compared to other protein coding counterparts.

LncRNAs are transcripts of longer than 200 bp.They have important roles in cellular processes like transcriptional regulation, chromosome remodeling, post-translational modifications and disruption in them may lead to disease conditions.

Colon cancer associated transcript-1 (CCAT1) is consistently upregulated in and is associated with pathogenesis of a number of malignancies, including gastric carcinoma, colon cancer, gallbladder cancer and hepatocellular carcinoma.

CCAT1 was identified initially in colon cancer Zhao (2016), who demonstrated that high expression of CCAT1 in CRC plasma may be used as predictive biomarker for screening of CRC.

The dysregulated expression of CCAT1 affects not only tumorigenesis, but also clinical manifestation, such as tumor size, lymph node metastasis, TNM stage, differentiation, invasion, patient survival and treatment outcome. This finding renders CCAT1 attractive as target for therapeutic intervention in cancer. The current available studies of the expression, clinical relevance, biological behavior and regulatory mechanism of CCAT1 in various cancers have been described. Also, the potential roles of CCAT1 in the diagnosis, prognostic evaluation and treatment of cancers have been discussed.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with colorectal cancer

Exclusion Criteria:

* 1. Patients with colorectal cancer that had been received chemotherapy, radiotherapy or surgical treatment.

  2. History of non-precancerous benign colorectal diseases (Irritable bowel syndrome, colitis, appendicitis, diverticulitis, paralytic ileus & intussusception).

  3. History of benign or malignant tumors in other organs.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: normal healthy individuals. precancerous colorectal diseases colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic value of long noncoding RNA (CCAT1) expression | baseline
  Evaluate the clinical utility of detecting long noncoding RNA (CCAT1) expression in diagnosis of colorectal cancer patients & its relation to tumor staging.

REFERENCES:
- [Background] Zhao B, Lu M, Wang D, Li H, He X. Genome-Wide Identification of Long Noncoding RNAs in Human Intervertebral Disc Degeneration by RNA Sequencing. Biomed Res Int. 2016;2016:3684875. doi: 10.1155/2016/3684875. Epub 2016 Dec 20. PMID 28097131